CLINICAL TRIAL: NCT00720902
Title: Assessment of Cardiovascular Risk Markers in GH Deficient Patients With Nonsecreting Pituitary Adenomas
Brief Title: Adult Growth Hormone Deficiency and Cardiovascular Risk
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Pamela U. Freda, Associate Professor of Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAB9681 (Serono-001); Serono-001 (Other: protocol)
Record Dates: First submitted 2008-06-16; First posted 2008-07-23 (Estimated); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth hormone
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Blood Specimen Collection; Growth Hormone-Releasing Hormone; Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A - Normal growth hormone secretion (Active Comparator): Patients who have undergone transsphenoidal surgery for a pituitary adenoma and have normal growth hormone secretion: Subjects will undergo a clinical exam with vital signs and blood draws, anthropometric measurements and skin fold thickness assessments. Subjects will also undergo GH stimulation testing with growth hormone releasing hormone (GHRH) & arginine, MRI and MR spectroscopy, carotid ultrasound, and have an endothelial cell biopsy.
  Interventions: Procedure: Blood draws; Drug: growth hormone releasing hormone (GHRH) & arginine; Procedure: Carotid ultrasound; Procedure: MRI; Procedure: Endothelial cell biopsy
- B - Growth hormone deficient (Active Comparator): Patients who have undergone transsphenoidal surgery for pituitary adenoma who are growth hormone deficient: Subjects will undergo a clinical exam with vital signs and blood draws, anthropometric measurements and skin fold thickness assessments. Subjects will also undergo GH stimulation testing with growth hormone releasing hormone (GHRH) & arginine, MRI and MR spectroscopy, carotid ultrasound, and have an endothelial cell biopsy.
  Interventions: Procedure: Blood draws; Drug: growth hormone releasing hormone (GHRH) & arginine; Procedure: Carotid ultrasound; Procedure: MRI; Procedure: Endothelial cell biopsy

INTERVENTIONS:
Procedure: Blood draws — Subjects will have serum cardiovascular markers assessed
Drug: growth hormone releasing hormone (GHRH) & arginine — Subjects will receive GHRH and arginine intravenously and then have blood drawn at frequent intervals over a 90 minutes to assess growth hormone secretion.
Procedure: Carotid ultrasound — Subjects will have an ultrasound of their neck to assess their carotid arteries to look for intima-medial thickness.
Procedure: MRI — Subjects will have MRI and MR spectroscopy of the abdomen and lower extremities to assess for fat in internal organs and muscle.
Procedure: Endothelial cell biopsy — Subjects will undergo endothelial cell biopsies to harvest endothelial cells to study. It will occur once and takes approximately 20 minutes. Patients will have an iv placed and then a sterile wire is passed back and forth in the iv a couple of times. Three wires are passed.

SUMMARY:
This protocol will assess the cardiovascular risk associated with growth hormone deficiency in adults. We will use multiple modalities to assess risk for heart attacks or strokes including blood work, ultrasound, MRI and endothelial cell biopsies in both patients who are growth hormone deficient and in patients with normal growth hormone secretion. We hypothesize that adults with growth hormone deficiency will have results suggestive of an increased risk for cardiovascular disease.

DETAILED DESCRIPTION:
Subjects will first be tested for possible growth hormone deficiency. This will be done by administering two intravenous medications that should stimulate growth hormone secretion and we will measure growth hormone in the blood every 30 minutes following the administration. Once we have the results on enough subjects we will split the cohort into those subjects who are growth hormone deficient and those who have normal growth hormone. The two groups will each undergo various tests all designed to assess some component of cardiovascular risk. Ultimately we will compare the results of each test to see if those who are growth hormone deficient have an increased risk for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 years or older who have undergone transsphenoidal surgery for a clinically non-secreting pituitary adenoma

Exclusion Criteria:

* Currently taking growth hormone, radiation therapy in the past 5 years, changes in dose of other pituitary hormone replacement therapy in past 3 months, taking hydrocortisone (or its equivalent) at a dose of > 30 mg/day, pregnant or nursing women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-02; Primary Completion 2010-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Ausiello, MD, Study Director — Columbia University
Locations (1):
- Columbia University, College of Physicians and Surgeons, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Growth Hormone (GH) Sufficient Participants: Participants with normal growth hormone secretion.
- Growth Hormone (GH) Deficient Participants: Participants with growth hormone secretion deficiency
Period: Overall Study
Arm/Group | Growth Hormone (GH) Sufficient Participants | Growth Hormone (GH) Deficient Participants
Started | 4 | 3
Completed | 0 | 3
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Unable to perform testing, lack of test agent and the Study terminated | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- GH Sufficient Participants: Participants with normal growth hormone secretion.
- GH Deficient Participants: Participants with growth hormone secretion deficiency.
- Total: Total of all reporting groups
Arm/Group | GH Sufficient Participants | GH Deficient Participants | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: C-reactive Protein (CRP) Levels
Description: C-reactive protein (CRP) levels in GH sufficient and GH deficient participants
Time Frame: Day 1
Population: Study was terminated early due to insufficient enrollment and lack of GHRH study medication to be administered. The medication became unavailable in the US after enrollment began, but before that testing could be performed. Without that testing, further classification of subjects as sufficient or deficient could not be performed and the remainder of the tests could not be done. Partial testing was only done on 3 GH deficient subjects and the results of this are reported.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 3
ng/dL |  | 14.46 (14.90)

2. Primary Outcome: Homocysteine Level
Description: Homocytsteine levels in GH sufficient and GH deficient participants
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 3
micromol/L |  | 8.04 (0.90)

3. Primary Outcome: Total Cholesterol Level
Description: Total cholesterol levels in GH sufficient and GH deficient participants
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 3
mg/dL |  | 271 (90.5)

4. Secondary Outcome: Percentage of Fat Measured by DXA DEXA
Description: Percentage of total body fat and trunk fat as measured by DXA
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 3
Percent
  Total body fat |  | 42.33333333 (8.73)
  Trunk fat |  | 21 (3.60)

5. Secondary Outcome: Lean Body Mass by DXA DEXA
Description: Lean body mass as measured by DXA
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 3
kg |  | 46.67 (2.89)

6. Secondary Outcome: Insulin Sensitivity as Assessed by Fasting Insulin Levels
Description: Insulin sensitivity as assessed by fasting insulin levels
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 3
mIU/L |  | 35.5 (28.94)

7. Secondary Outcome: Glucose Levels as Assessed by an Oral Glucose Tolerance Test
Description: Glucose levels as assessed by an oral glucose tolerance test
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 3
mg/dL |  | 91.33 (4.163)

8. Secondary Outcome: Endothelial Function as Assessed by Flow Mediated Dilatation and Endothelial Cell Biopsy
Description: Endothelial function as assessed by flow mediated dilatation and endothelial cell biopsy for measurement of inflammatory markers.
Time Frame: Day 1
Population: Study was terminated early due to insufficient enrollment and lack of GHRH study medication to be administered. The medication became unavailable in the US after enrollment began, but before that testing could be performed. Without that testing, further classification of participants as sufficient or deficient could not be performed and the remainder of the tests could not be done. As a result, data were not collected for GH sufficient or GH deficient participants for this outcome measure
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Carotid Intimal-medial Thickness Studies as Assessed by Ultrasound
Description: Carotid intimal-medial thickness studies will be measured by ultrasound
Time Frame: Year 1
Population: Study was terminated early due to insufficient enrollment and lack of GHRH study medication to be administered. The medication became unavailable in the US after enrollment began, but before that testing could be performed. Without that testing, further classification of participants as sufficient or deficient could not be performed and the remainder of the tests could not be done. As a result, data were not collected for GH sufficient and GH deficient participants.
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Intramyocellular Lipid Content Using MRI and MR Spectroscopy
Description: Intramyocellular lipid content using MRI and MR spectroscopy of the soleus muscle was performed.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent water signal
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 3
Percent water signal |  | 0.011763 (0.00159)

11. Secondary Outcome: Intrahepatic Lipid Content Using MRI and MR Spectroscopy
Description: Intrahepatic lipid (IHL) content using MRI and MR spectroscopy of the liver was performed.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent water signal
Arm/Group | GH Sufficient Participants | GH Deficient Participants
Number analyzed (Participants) | 0 | 3
Percent water signal |  | 9.97 (7.17)

ADVERSE EVENTS:
Groups:
- GH Sufficient Participants: Participants with a history of pituitary disease, but who have a history of being GH sufficient.
- GH Deficient Participants: Participants with a history of pituitary disease who have a history of being GH deficient
Arm/Group | GH Sufficient Participants | GH Deficient Participants
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes